CLINICAL TRIAL: NCT00671528
Title: Double-blind Evaluation of the Safety and Efficacy of Quadriderme® (Betamethasone Diproprionate, Clotrimazole and Gentamicin) Compared With Betamethasone Diproprionate Combined With Gentamicin Sulfate and With Betamethasone Diproprionate in the Treatment of Impetiginous Eczema
Brief Title: Safety and Efficacy of Quadriderme® in the Treatment of Impetiginous Eczema (Study P05134AM4)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: terminated early due to lack of recruitment [only 3 of 207 subjects were enrolled]
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05134; EudraCT No.: 2007-004980-23
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Results first posted 2011-06-16 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Dermatitis, Atopic; Eczema, Atopic; Skin Diseases, Eczematous
Keywords: Impetiginous
MeSH Terms: conditions — Dermatitis, Atopic; Skin Diseases, Eczematous | interventions — Clotrimazole; Gentamicins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- QUADRIDERME® cream (Experimental): QUADRIDERME® cream (betamethasone diproprionate, clotrimazole, and gentamicin sulfate)
  Interventions: Drug: Cream (betamethasone diproprionate, clotrimazole, and gentamicin sulfate)
- Betamethasone and Gentamicin (Active Comparator): Combination of betamethasone diproprionate cream and gentamicin sulfate cream
  Interventions: Drug: Cream (betamethasone diproprionate and gentamicin)
- Betamethasone (Active Comparator): Betamethasone diproprionate cream
  Interventions: Drug: Cream (betamethasone diproprionate)

INTERVENTIONS:
Drug: Cream (betamethasone diproprionate, clotrimazole, and gentamicin sulfate) — Betamethasone diproprionate 0.05%, clotrimazole 1%, and gentamicin sulfate 0.1% cream applied in a thin layer that covers the affected and surrounding area 2 times a day (BID), morning and night for a maximum period of 28 days or until 5 days after total remission of the signs and symptoms, but never more than 28 days.
  Other Names: QUADRIDERME® cream, SCH 000411
  Arms: QUADRIDERME® cream
Drug: Cream (betamethasone diproprionate and gentamicin) — Betamethasone diproprionate 0.05% and gentamicin sulfate 0.1% cream applied in a thin layer that covers the affected and surrounding area BID, morning and night for a maximum period of 28 days or until 5 days after total remission of the signs and symptoms, but never more than 28 days.
  Arms: Betamethasone and Gentamicin
Drug: Cream (betamethasone diproprionate) — Betamethasone diproprionate 0.05% cream applied in a thin layer that covers the affected and surrounding area BID, morning and night for a maximum period of 28 days or until 5 days after total remission of the signs and symptoms, but never more than 28 days.
  Arms: Betamethasone

SUMMARY:
This is a parallel-group, randomized, active-controlled, double-blind, Phase 4 trial comparing three creams in the treatment of impetiginous eczema:

* Arm A: QUADRIDERME® cream (betamethasone diproprionate, clotrimazole, and gentamicin sulfate)
* Arm B: Combination of betamethasone diproprionate cream and gentamicin sulfate cream
* Arm C: Betamethasone diproprionate cream

At 7 sites, in Portugal, a total of 207 subjects will be randomized using a 1:1:1 randomization ratio to receive one of the three possible treatments for a maximum period of 28 days or until 5 days after total remission of the signs and symptoms, but never more than 28 days. Assessments will be made of level of improvement of the target area in each treatment group, number of days for total remission, and safety profile.

Note: This study was terminated early due to lack of recruitment (only 3 of the 207 planned participants were enrolled). Statistical analyses were not performed.

Further, 7 sites were planned, but only 4 sites were approved out of which 3 sites were initiated.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age: 12 years
* Good general health confirmed by clinical history and a physical and skin examination (excluding area of skin with impetiginous eczema).
* Diagnosis of impetiginous eczema.
* Ability to understand the procedures of the protocol and follow the requirements during the course of the study.
* Results of routine laboratory tests - hemogram with leukogram and platelet count, creatinine, glucose, sed. rate, IgE level and transaminases; along with plasma cortisol and adrenocorticotropic hormone (ACTH) levels prior to the start of the treatment. These results must all be within normal limits or not clinically relevant in order to be included in the trial.

Exclusion Criteria:

* Pregnant participants or women of childbearing age who are not using birth control methods considered reliable by the attending physician.
* Participants with a history of hypersensitivity to any of the components of the medication being studied.
* Participants in whom the extent or severity of the lesions requires treatment of a different type than what is planned for this trial.
* Participants who need any other type of topical or systemic medication during the trial that might affect the course of the disease.
* Participants who have been treated with other topical medications during the 14-day period prior to the start of the trial.
* Participants who have received systemic corticosteroids or any other immunosuppressant medication during the 28-day period prior to the start of the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to lack of recruitment, the study was terminated early. Only 3 participants of the anticipated 207 participants were enrolled.
Groups:
- Quadriderme® Cream: Combination of Betamethasone diproprionate 0.05%, clotrimazole 1%, and gentamicin sulfate 0.1% applied in a thin layer that covers the affected and surrounding area 2 times a day (BID), morning and night for a maximum period of 28 days or until 5 days after total remission of the signs and symptoms, but never more than 28 days.
- Betamethasone Diproprionate and Gentamicin Sulfate Cream: Combination of Betamethasone diproprionate 0.05% cream and gentamicin sulfate 0.1% applied in a thin layer that covers the affected and surrounding area BID, morning and night for a maximum period of 28 days or until 5 days after total remission of the signs and symptoms, but never more than 28 days.
- Betamethasone Diproprionate Cream: Betamethasone diproprionate 0.05% cream applied in a thin layer that covers the affected and surrounding area BID, morning and night for a maximum period of 28 days or until 5 days after total remission of the signs and symptoms, but never more than 28 days.
Period: Overall Study
Arm/Group | Quadriderme® Cream | Betamethasone Diproprionate and Gentamicin Sulfate Cream | Betamethasone Diproprionate Cream
Started | 1 | 1 | 1
Completed | 1 | 1 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quadriderme® Cream | Betamethasone Diproprionate and Gentamicin Sulfate Cream | Betamethasone Diproprionate Cream | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 0 | 0 | 1 | 1
  >=65 years | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Improvement of Individually Measured Signs of the Disease
Description: Percent improvement of individually measured signs of the disease (erythema, vesiculation, scaling, pruritis) in a given target area that was chosen by the investigator was assessed objectively & quantified on a scale of 0-5 (0-absent, 5-very intense). Overall assessment reflected the changes in the disease & was carried out by the investigator.
  The following scale was used:
  1. Cure- Complete remission
  2. > 75% reduction: Marked improvement
  3. 50-75% reduction: Moderate improvement
  4. 25-50% reduction: Slight improvement
  5. <25% reduction: Ineffectiveness
  6. Worsening of signs & symptoms
Time Frame: Days 1 (prior to start of treatment), 8, 15, 21, and 28.
Population: Due to lack of participant recruitment and therefore study termination, no analyses were performed.
Arm/Group | Quadriderme® Cream | Betamethasone Diproprionate and Gentamicin Sulfate Cream | Betamethasone Diproprionate Cream
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Number of Days Required to Achieve Total Remission
Description: The speed of action, measured as the number of days required to achieve total remission of all signs and symptoms of the disease.
Time Frame: Up to 28 days
Measure: Number; unit: Days
Arm/Group | Quadriderme® Cream | Betamethasone Diproprionate and Gentamicin Sulfate Cream | Betamethasone Diproprionate Cream
Number analyzed (Participants) | 1 | 1 | 1
Days | 15 | 15 | 8

ADVERSE EVENTS:
Arm/Group | Quadriderme® Cream | Betamethasone Diproprionate and Gentamicin Sulfate Cream | Betamethasone Diproprionate Cream
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
This study was terminated early due to lack of recruitment (only 3 of 201 participants were enrolled). Statistical analyses were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigators agree not to publish or publicly present any interim results of the study without prior written consent of the SPONSOR. The principal investigator further agrees to provide 45 days written notice to the sponsor prior to submission for publication or presentation to permit the SPONSOR to review copies of abstracts or manuscripts for publication which report any results of the study. The SPONSOR shall have the right to review and comment on any presentation.